CLINICAL TRIAL: NCT02067624
Title: Effects of Thai Massage on Patients With Wrist Extensor Muscles Latent Myofascial Trigger Points
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mae Fah Luang University Hospital (Other)
Responsible Party: Principal Investigator, Dr. Vitsarut Buttagat, Head of School of physical Therapy, Mae Fah Luang University, Mae Fah Luang University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 55218152-4
Record Dates: First submitted 2014-02-18; First posted 2014-02-20 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Patients With Latent Myofascial Trigger Point
MeSH Terms: interventions — Medicine, Thai Traditional

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thai massage (Experimental): The participants will receive a thirty minutes session of Thai massage onto the wrist extensor groups muscle for 9 sessions
  Interventions: Other: Thai massage
- Sham Ultrasound therapy (Sham Comparator): The participants will receive a thirty minutes session of sham ultrasound therapy onto the wrist extensor groups muscle for 9 sessions
  Interventions: Other: Thai massage

INTERVENTIONS:
Other: Thai massage

SUMMARY:
The purpose of this study was to investigate the effect of Thai massage on pressure pain threshold, pain intensity, wrist range of motion, grip strength and patient satisfaction in patients with wrist extensor muscles latent Myofascial trigger points.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age between 18 - 40 years old
* The participants have at least one latent trigger point in the wrist extensor groups muscles.
* The participants will be able to follow instructions.
* Good communication and cooperation.

Exclusion Criteria:

* Contraindications of traditional Thai massage
* Tennis elbow or Golf's elbow
* Poor skin sentation

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2014-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Pressure Pain Threshold as a measure by algometry | 5 weeks

SECONDARY OUTCOMES:
Pain scores on visual analog scale | 5 weeks
Wrist Range of motion as a Measure by goniometer | 5 weeks
Grip strength as a measure by hand-held dynamometer | 5 weeks
Patient satisfaction level | 5 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- School of Health Science, Mae Fah Luang University, Mueang, Changwat Chiang Rai, Thailand

REFERENCES:
- [Derived] Buttagat V, Kluayhomthong S, Areeudomwong P. The beneficial effects of traditional Thai massage on young patients with latent myofascial trigger points in the wrist extensor muscles: A randomized controlled trial. J Bodyw Mov Ther. 2024 Oct;40:1201-1207. doi: 10.1016/j.jbmt.2023.04.024. Epub 2023 Apr 13. PMID 39593435